CLINICAL TRIAL: NCT05842239
Title: Hyperbaric Oxygen Therapy for Men Suffering From Infertility Due to Oligospermia: a Pilot Study
Brief Title: Hyperbaric Oxygen Therapy for Men Suffering From Infertility Due to Oligospermia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 209-22-ASF
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Oligospermia
MeSH Terms: conditions — Oligospermia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperbaric Oxygen Therapy active arm (Experimental): The protocol comprises of 60 consecutive hyperbaric oxygen treatment (HBOT) sessions, 5 sessions per week within a three months' period.
  Interventions: Device: Hyperbaric oxygen therapy

INTERVENTIONS:
Device: Hyperbaric oxygen therapy — Each session will include exposure of 90 minutes to 100% at 2 ATA, with 5 minutes air breaks every 20 minutes

SUMMARY:
Infertility in a couple is defined as the inability to achieve conception despite one year of frequent, unprotected intercourse. Infertility affects approximately 12% of couples attempting to conceive. The goal of this study is to explore the potential beneficial effect of HBOT on sperm count of infertile male due to oligospermia.

DETAILED DESCRIPTION:
Infertility in a couple is defined as the inability to achieve conception despite one year of frequent, unprotected intercourse. Infertility affects approximately 12% of couples attempting to conceive. The male factor is equally attribute to couple infertility like woman infertility.

Male infertil¬ity may have many reasons. In up to 90% of male infertility cases, there is a decrease in sperm count or the might show poor sperm quality. During spermatogenesis, mitochondria undergo continuous morphological and distributional changes with germ cell development. Deficiencies in these processes lead to mitochondrial dysfunction and abnormal spermatogenesis, thereby causing male infertility.

In addition to mitochondria, telomer also play a significant role in sperm functionality. Telomere length is considered one of the most relevant biological markers of genomic stability. The negative impact of telomere shortening on sperm quality has been suggested as an important indicator of male infertility.

It is now understood that Hyperbaric oxygen treatment (HBOT), triggers both oxygen and pressure sensitive genes, resulting in inducing mitochondrial proliferation, increase in complex I activity and those mitochondrial efficiency. With respect to telomers, in a recent study, it was demonstrated that HBOT can induce telomeres elongation.

The goal of this study is to explore the potential beneficial effect of HBOT on sperm count of infertile male due to oligospermia.

All eligible participants will receive hyperbaric treatment. The treatment will be administrated in a multi-place chamber. The protocol comprises of 60 daily sessions, 5 sessions per week within a three-month period. Each session includes breathing 100% oxygen by mask at 2ATA for 90 minutes with 5-minute air breaks every 20 minutes.

The evaluation procedure will be performed 4 times, at baseline, after 40 sessions, end of the treatment period and 60 days after the treatment ended, and includes sperm analysis, sperm and lymphocyt telomeres length.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 21 years
2. At least two sperm examination showing oligospermia (<15·106 sperm/mL)
3. Diagnosis of idiopathic oligospermia.
4. Subject willing and able to read, understand and sign an informed consent

Exclusion Criteria:

1. Inability to attend scheduled clinic visits and/or comply with the study protocol
2. Active malignancy
3. Previous treatment with chemotherapy and/or radiation therapy
4. Substance use at baseline
5. Severe or unstable physical disorders or major cognitive deficits at baseline
6. HBOT for any reason prior to study enrolment
7. Chest pathology incompatible with pressure changes (including moderate to severe asthma)
8. Ear or Sinus pathology incompatible with pressure changes
9. Chronic disease like diabetes mellitus, ischemic heart disease etc.
10. Active smoking

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sperm count | At baseline, 3 months
  Change from baseline in sperm count measured by Sperm Analysis

SECONDARY OUTCOMES:
Sperm morphology | At baseline, 3 months, 9 months
  Change from baseline in sperm morphology measured by Sperm Analysis
Sperm count | 9 months
  Change from baseline in sperm count measured by Sperm Analysis
Sperm motility | At baseline, 3 months, 9 months
  Change from baseline in sperm motility measured by Sperm Analysis
Sperm telomeres length | At baseline, 3 months, 9 months
  Change from baseline in sperm telomeres length
Lymphocyte telomeres length | At baseline, 3 months, 9 months
  Change from baseline of lymphocyte telomeres length

OTHER OUTCOMES:
Change from baseline of anaerobic threshold by cardio-pulmonary exercise testing CPET | At baseline, 3 months
  CPET determines the anaerobic threshold that is expected to change through the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Shachar Finci, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- The Sagol Center for Hyperbaric Medicine and Research Shamir Medical Center (Assaf Harofeh), Ẕerifin, Israel